CLINICAL TRIAL: NCT06184984
Title: Metabolic Availability of Methionine in Monggo Meal Among Women of Reproductive Age Using Indicator Amino Acid Oxidation (IAAO)
Brief Title: Metabolic Availability of Methionine in Mung Beans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Nutrition Research Institute, Philippines (Other Government)
Collaborators: International Atomic Energy Agency (Other Government); Mahidol University (Other)
Responsible Party: Principal Investigator, Johanne B. Guilaran, Principal Investigator, Food and Nutrition Research Institute, Philippines
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FIERC-2024-030
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-10

CONDITIONS: Healthy Women of Child Bearing Potential
Keywords: Metabolic Availability; Methionine; IAAO; Mung beans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methionine metabolic availability in mung beans (Experimental): Participants will be seen initially for pre-study assessment. They will then be studied for up to 7 times.
  The participants will be expected to participate in 7 different sets of experiments which will take 2 to 3 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein free-cookies and/or cooked mung bean, which will be provided by the investigators.
  Interventions: Dietary Supplement: Metabolic availability of methionine in mung beans

INTERVENTIONS:
Dietary Supplement: Metabolic availability of methionine in mung beans — Each participant will randomly receive 7 different levels of methionine provided as free amino acids and cooked mung beans.

SUMMARY:
The goal of this study is to determine the protein quality of Philippine mung beans. The main objective of this study is to determine the metabolic availability of methionine in mung beans that the body can use. We will test the mung beans by studying them after cooking them as sauté.

This research is being done in order to bridge the gap between knowledge of protein requirement and the amount of food needed to meet that requirement. Results from this study will be important for recommendations guiding food choices of mung beans as a major protein source in the diet.

Each study participant will be part of seven (7) different experimental diets, and randomly assigned to one of the diets every time. Four (4) reference diets would be based on egg protein composition, and three (3) test diets will have protein from cooked mung beans.

Each experimental diet will be studied over 3 days: 2 adaptation days and 1 study day. The meals during the 2-day adaptation period would be consumed at home. On the study day, following a 10 to 12-h overnight fast, the study participants will come to the research unit at the Department of Science - Food and Nutrition Research Institute (DOST-FNRI), Gen. Santos Ave., Bicutan, Taguig City, Philippines, for a period of 8 to 9 hours and consume the diets as 9 hourly meals.

DETAILED DESCRIPTION:
The pre-study assessments will include the measurement of Basal Metabolic Rate (BMR) / Resting Energy Expenditure (REE) by open-circuit indirect calorimetry, and body composition (fat and fat-free mass) by deuterium oxide dilution technique.

The study protocol is a 3-day experimental protocol (2 days of adaptation plus 1 study day), with an interval of ≥1 week to ensure complete tracer washout.

Each participant is adapted to the test diets for two days to provide them with adequate energy and protein (isonitrogenous diet), and to stabilize their metabolic pool. The energy during the adaptation period is provided at resting energy expenditure (REE/BMR) x 1.7 and protein 1.0 g.kg-1.d-1. During this period, each participant will be expected to consume 4 meals per day consisting of a protein liquid drink and protein free-cookies and/or cooked mung bean meal, which the investigators will provide.

On the study day, after a 10-12 h overnight fast, the participants will come to the research unit for 8-9 h, and receive 9 isonitrogenous, isocaloric hourly meals, each representing one-tenth of the participant's total daily protein (1 g.kg-1.d-1) and energy requirement (1.5 x REE/BMR).

The protein is supplied either as the reference amino acid mixture or as a combination of the reference amino acid mixture and the test proteins. The amount of each test protein provided at each level of selected IAA (Indispensable Amino Acid) intake should be calculated based on the concentration from all sources.

Indicator AA (Amino Acid), phenylalanine is provided at 30 mg.kg-1.d -1 in all study diets (from food protein and isotope). The amount of phenylalanine provided from crystalline amino acid should be deducted depending on the natural phenylalanine content in the test protein.

The non-protein energy in the test diets is provided through a flavored sugar-oil drink and protein-free wheat starch cookies.

The reference amino acid mixture, non-labelled crystalline phenylalanine, tyrosine, and selected IAA are added and mixed with the sugar-oil drink before administering the hourly mini-meals. The test proteins are separately administered to the participants with each mini-meal.

Breath samples are collected before starting the first mini meal, at baseline (before the tracer protocol; a stable fed state in breath 13CO2 background abundance occurs after 4 hourly mini-meals) and every 15-min during isotopic steady state (approximately 2.5 h after starting the isotope). Three breath samples should be collected in 10 mL non-silicon-coated tubes using a collection mechanism that permits the removal of dead-space air at each time point. When breath collection coincides with an hourly meal, the breath sample should be collected first, followed by the meal. Then, all breath samples are stored at room temperature, pending analysis.

Enrichment of 13C in breath is analyzed by continuous flow isotope ratio mass spectrometer. The 13CO2 enrichment in the breath samples due to isotopic administration during the fed state is expressed as atom % excess (APE) over baseline. Then, the fraction of 13CO2 (F13CO2) from the tracer phenylalanine oxidation in relation to the amount administered is calculated.

The reference and test IAAO response slopes are calculated from F13CO2 measurements and the respective IAA intakes using a linear mixed effect regression mode, with a common origin of F13CO2 response at base test IAA intake. The metabolic availability (MA) of test amino acid in the test meal is determined by the slope-ratio method using the following equation:

MA (%) = (Test protein slope × 100)/ Reference slope

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant
2. Non-lactating
3. Stable body weight
4. Healthy, with no known clinical condition that would affect protein or AA metabolism, e.g. Diabetes
5. Not on any medications that could affect protein or amino acid metabolism e.g. steroids.

Exclusion Criteria:

1. Unwillingness to participate or unable to tolerate the diet
2. Recent history of weight loss within the last 3 months or on a weight-reducing diet
3. Inability to tolerate study diets (e.g. Allergy to ingredients)

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Metabolic availability of methionine in mung beans | 2 years
  Protein quality of mung beans measured as metabolic availability using the IAAO method

CONTACTS AND LOCATIONS:
Overall Officials: Johanne B Guilaran, Bachelor's, Principal Investigator — Department of Science and Technology - Food and Nutrition Research Institute
Locations (1):
- Department of Science and Technology - Food and Nutrition Research Institute, City of Taguig, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No